CLINICAL TRIAL: NCT05563818
Title: Monitoring Symptoms Severity in Arabic Speaking Schizophrenic Patients Using Mobile Phone Speech Analysis: A Proof-of-Concept Study
Brief Title: Using Speech to Monitor Symptom Severity in Arabic Speaking Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Collaborators: Winterlight Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: HIK-WL-SCZ-2021-01
Record Dates: First submitted 2022-03-08; First posted 2022-10-03 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Schizophrenic Disorders; Mental Disorders; Speech; Voice; Language; Natural Language Processing; Behavioral Symptoms
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Speech; Language; Behavioral Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arabic-speaking individuals with schizophrenia: Approximately 56-60 Arabic-speaking individuals with a DSM-5 diagnosis of schizophrenia
  Interventions: Other: WinterLight Mobile Phone Speech Analysis

INTERVENTIONS:
Other: WinterLight Mobile Phone Speech Analysis — N/A- observational study

SUMMARY:
Brief Summary:

Definition: A short description of the clinical study, including a brief statement of the clinical study's hypothesis, written in language intended for the lay public.

Limit: 5000 characters. The purpose of this study is to investigate the relationship between speech features and severity of positive and negative clinical symptoms in Arabic speaking patients with schizophrenia. Individuals will be invited to participate in this study because (1) they have a confirmed clinical diagnosis of schizophrenia; (2) they plan to receive routine clinical care for schizophrenia at one of the four participating sites; (3) they speak Arabic as a first language.

Participants must be between the ages of 18-65 years. Participation will involve seven visits consisting of one baseline visit and six monthly follow-up visits. All participants will continue to receive routine clinical care.

Participation in this research will involve providing speech samples using standardized tasks collected using an electronic device. Additionally, study team members will assess positive and negative symptoms of schizophrenia using validated questionnaires.

DETAILED DESCRIPTION:
Speech disorganization is a key feature of schizophrenia. The development of computerized tools to assess speech disorganization is rapidly growing in schizophrenia research. Several early studies showed that changes in speech distinguish schizophrenia patients from healthy controls and assist in differential diagnostics and relapse prevention (1). The Winterlight app can be used for speech collection and assessment and uses speech-based artificial intelligence to identify vocal biomarkers capable of detecting changes in cognitive/clinical symptoms.

Symptom rating scales remain the primary mode of assessing the nature and severity of schizophrenia and the magnitude of any change over time. The Positive and Negative Symptom Scale (PANSS) is a 30-item rating scale that was developed to measure the symptom severity of patients with schizophrenia and assess their dimensions (2). It has been widely used in clinical trials of schizophrenia and is considered as the "gold standard" for the assessment of antipsychotic treatment efficacy.

The goal of this study is to test the hypothesis that quantitative measures derived from speech samples acquired using the Winterlight application will be associated with positive and negative symptom subscores as assessed by the PANSS.

The investigators will use speech-based artificial intelligence methods to identify aspects of voice and language that are related to schizophrenia symptoms in Arabic-speaking patients.

Data collected may be used to evaluate:

1. The relationship between speech measures and PANSS subscores at baseline.
2. The relationship between changes in speech measures and changes in positive symptoms over time.
3. The relationship between changes in speech measures and changes in negative symptoms over time.
4. The ability for speech measures to be used to predict psychotic relapse in individuals with schizophrenia.
5. The feasibility of predicting relapse based on speech and sociodemographic variables.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 65 years
2. Confirmed clinical diagnosis of schizophrenia as per the DSM-5 criteria, at any stage of disease.
3. Planned to receive routine clinical care for schizophrenia in the study site for the next 6 months.
4. Arabic is first language

Exclusion Criteria:

1. Illiterate.
2. Catatonic schizophrenia subtype.
3. Neurological disorder or major health problem.
4. Severe substance use disorder using DSM-5 criteria.
5. Risk to self or others.
6. Patient with any speech disorder or treated/planned to be treated with any medication known to impact speech (e.g. first-generation antipsychotics)
7. Patient or family member is unable to provide consent to participate in the study.
8. Participation in another clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from four medical sites in the Middle East North Africa (MENA) region, which are located in Jordan, Saudi Arabia, Egypt, and Algeria.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Speech features derived from the Winterlight Assessment (WLA). | up to month 6
  Acoustic and linguistic measures of speech acquired using the Winterlight Application
Positive and Negative Syndrome Scale (PANSS) including total score, positive subscore, negative subscore and psychopathology subscore. | up to month 6
  30-item clinical scale to assess positive and negative symptoms severity in people with schizophrenia.

SECONDARY OUTCOMES:
Change in speech features derived from the Winterlight Assessment (WLA). | Change from baseline to month 6
  Baseline to endpoint (6 month) change on acoustic and linguistic measures of speech computed based on the WLA.
Change in Positive and Negative Syndrome Scale (PANSS) including total score, positive subscore, negative subscore and psychopathology subscore. score measured by the PANSS positive sub-score | Change from baseline to month 6
  Baseline to endpoint (6 month) change on 30-item clinical scale to assess positive and negative symptoms severity in people with schizophrenia
Incidence of psychotic relapse | Change from baseline to month 6
  Psychotic relapse is defined as: hospitalization, suicidal/homicidal ideation, violent behavior, a 25% increase in the PANSS total score, or a significant increase in at least one of several pre-specified PANSS items.

CONTACTS AND LOCATIONS:
Locations (4):
- Mustapha University Hospital, Algiers, Algeria
- Ain Shams Hospital, Cairo, Egypt
- Mental Health Hub, Amman, Jordan
- Jeddah Psychiatry Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Boer JN, Brederoo SG, Voppel AE, Sommer IEC. Anomalies in language as a biomarker for schizophrenia. Curr Opin Psychiatry. 2020 May;33(3):212-218. doi: 10.1097/YCO.0000000000000595. PMID 32049766
- [Background] Kay SR, Fiszbein A, Opler LA. The positive and negative syndrome scale (PANSS) for schizophrenia. Schizophr Bull. 1987;13(2):261-76. doi: 10.1093/schbul/13.2.261. PMID 3616518